CLINICAL TRIAL: NCT06432426
Title: The Effect of Virtual Exercise on Elderly Breast Cancer Survivors on Functionality, Muscular Strength, and Quality of Life Effecto-B):
Brief Title: Virtual Exercise on Elderly Breast Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 38330628
Record Dates: First submitted 2024-05-09; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer
Keywords: breast neoplasm; elderly; physical exercise; virtual reality
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Training Group (Experimental): Participants will undergo a postural balance rehabilitation program, utilizing a probed protocol for the elderly population with virtual reality via the Nintendo Wii Fit® and its peripheral Balance Board system. Supervised group sessions will be conducted twice a week for 9 weeks.
  Interventions: Behavioral: Virtual reality training group
- Standard physical exercise Group (Active Comparator): Participants will undergo a standardized physical exercise program based on a validated protocol designed for elderly breast cancer survivors
  Interventions: Behavioral: Standard physical exercise group

INTERVENTIONS:
Behavioral: Virtual reality training group — Participants will be given virtual reality games on Nintendo Wii Fit® and its peripheral Balance Board system. This equipment offers safe and engaging training protocols. Additionally, it ensures physical exercise in the three planes of movement (sagittal, frontal, and transverse) and with three difficulty levels, thus providing a linear progressive demand.
  Arms: Virtual Reality Training Group
Behavioral: Standard physical exercise group — Participants will be submitted to a standard physical exercise program based on the ACSM guidelines. Resistance training will involve exercises for arms and legs, using bodyweight self-loading and external weights. Balance exercises will include the three planes of movement.
  Arms: Standard physical exercise Group

SUMMARY:
Breast cancer (BC) is the most common neoplasia. Frequent for women and half of the new cases occur in people over 65 years of age. The treatment of BC generates adverse effects that deteriorate the physical functionality, muscle strength and quality of life of the survivors. This is more noticeable in elderly BC survivors. Physical exercise improves some adverse effects of BC, but few studies have focused on physical functionality, especially in older people. The elderly population reports the lowest adherence and lower level of physical activity. It is relevant to explore innovative and specific proposals for physical exercise for elderly survivors of BC. One solution may be virtual reality game-based exercise, which has been shown in healthy older people to significantly improve physical functionality and adherence compared to traditional physical exercise. The objective of our study is to estimate the feasibility and effect of a virtual reality-based exercise program on the functionality, muscle strength, and quality of life of older BC survivors, compared to a group undergoing traditional physical exercise.

DETAILED DESCRIPTION:
This is a randomized controlled study. It will be conducted at the Dr. Sotero del Río Assistance Complex, which receives Southeast Metropolitan Health Service patients. Participants: 60 women over 60yrs who completed their antineoplastic treatment at least two years ago will be recruited.

Functionality will be measured using the Short Physical Performance Battery (SPPB), which is specific for older individuals. Hydraulic Dynamometry (Jamar © hydraulic hand dynamometer) will evaluate isometric upper limb muscle strength. Quality of life shall be assessed using the EORTC QLQ C30 Quality of Life Questionnaire - with its EORTC QLQ-ELD14 module, validated in the Chilean population. Feasibility will be measured using recruitment rate (≥50%), retention rate (≥ 80%), adherence rate (75% of total sessions ≥14 sessions), and incidence of adverse events.

Candidates will be randomly assigned to either virtual reality or traditional exercise groups. Both training groups will involve supervised sessions twice a week for nine weeks. The traditional exercise group exercises will be for arms and legs, involving body weight and external weights. Meanwhile, the virtual reality group will follow a physical exercise protocol using the "Nintendo Wii Fit" console. After the 9th week, participants will be evaluated one month after completing the training program.

ELIGIBILITY:
Inclusion Criteria:

* Women between 60 and 80 years old.
* Diagnosis of primary breast carcinoma.
* Treated with at least two of the following treatments: surgery, radiotherapy, chemotherapy, hormone therapy, biological therapy.
* Minimum of 2 years and a maximum of 10 years after finishing treatments (surgery, chemotherapy, and radiotherapy).
* Being able to walk at least 4 meters independently or with a cane as assistive technology

Exclusion Criteria:

* Stage IV breast cancer.
* Previous cancer treatment for any type of cancer other than breast cancer (chemotherapy, radiotherapy, or endocrine therapy).
* Cognitive impairment measured by the abbreviated Mini-Mental State Examination with a score < 13 points.
* Medical contraindication to perform physical exercise.
* Self-reported of physical activity equivalent to the recent American College of Sports Medicine Exercise Guidelines for Cancer Patients and Survivors (150 min/week of moderate aerobic exercise and strength exercise twice a week).
* Body mass index < 18.5 kg/m2 or > 40 kg/m2.

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in the functionality | Baseline, week 9 and week 13
  Functionality will be measured by the Short Physical Performance Battery (SPPB). This battery is specific for older individuals and assess balance, walking speed, and lower extremity strength/endurance. It is a tool with moderate to excellent validity and excellent test-retest reliability (ICC=0.91).

SECONDARY OUTCOMES:
Change in upper limb muscle strength | Baseline, week 9 and week 13
  Upper body muscle strength will be assessed by manual grip strength measured with a hydraulic dynamometer (Jamar© hydraulic hand dynamometer) in kilograms. It is considered the gold standard for quantitative and objective evaluation of isometric hand and forearm muscle strength.
Change in lower limb muscle strength | Baseline, week 9 and week 13
  Lower body muscle strength will be measured using the 30-second Chair Stand Test. It has excellent validity and reliability in older adults. It is measured in the number of repetitions. The number of times the person can stand up from the chair in 30 seconds is recorded.
Change in the quality of life score | Baseline, week 9 and week 13
  Quality if life will be assessed with the QLQ C-30 questionnaire and the specific module QLQ-ELD14. The questionnaire could be self-administered and is validated to assess health-related quality of life in breast cancer patients. It has been validated in Spanish and in the Chilean population. Better quality of life is defined by a higher score (0-100) for global health status or overall quality of life.
Feasibility assesment | Baseline, week 1-9 and week 13
  It will be measured by the recruitment rate (>50%), retention rate (>80%), adherence rate (75% of total sessions >14 sessions), and the incidence of adverse effects. The measurements will be reported together as feasibility

CONTACTS AND LOCATIONS:
Overall Officials: Karol Ramírez-Parada, PT, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Complejo Asistencial Dr. Sótero del Río, Santiago, Puente Alto, Chile